CLINICAL TRIAL: NCT07224932
Title: A Randomized, Double-blind, Placebo-controlled Parallel Study of the Tolerability and Efficacy of High Cannabidiol (CBD) Cannabis Extract for the Treatment of Patients With Idiopathic Restless Legs Syndrome (RLS)
Brief Title: Tolerability and Efficacy of CBD Extract for RLS Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: BRC Therapeutics (Unknown); Biopharmaceutical Research Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-0682
Record Dates: First submitted 2025-10-06; First posted 2025-11-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Restless Leg Syndrome
Keywords: Restless Leg Syndrome; cannabis; BRC-002
MeSH Terms: conditions — Restless Legs Syndrome; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Half of the patients will be randomized to receive placebo orally. It is an oral solution of mono-, di-, and triglycerides
  Interventions: Drug: Placecbo
- BRC-002 (Experimental): Half of patients will be randomized to receive oral investigational product. BRC-002 is a non-scheduled high cannabidiol cannabis extract (<0.3% THC). The cannabinoids in BRC-002 are naturally biosynthesized within the Cannabis sativa L. plant.
  Interventions: Drug: BRC-002

INTERVENTIONS:
Drug: BRC-002 — BRC-002 is a non-scheduled cannabidiol (CBD) formulation (<0.3% THC). The cannabinoids in BRC-002 are naturally biosynthesized within the Cannabis sativa L. plant. BRC-002 is a high Cannabidiol Botanical extract (100 mg/mL).
  Other Names: Cannabidiol Formulation
  Arms: BRC-002
Drug: Placecbo — Oral solution of mono-, di-, and triglycerides
  Arms: Placebo Comparator

SUMMARY:
This study plans to learn more about the safety and tolerability of high Cannabidiol (CBD) cannabis extract (BRC-002) for use in Idiopathic Restless Legs Syndrome. Symptoms and side effects experienced while taking the study drug will be tracked to determine if this medication is safe to use.

DETAILED DESCRIPTION:
This randomized, placebo-controlled clinical trial will evaluate the safety, tolerability, and therapeutic effects of a high-CBD botanical extract in patients with idiopathic RLS. The study will examine changes in symptom severity, sleep quality, mood, and daily functioning to determine whether cannabinoid-based therapy offers a viable alternative or adjunctive treatment for RLS. Some inclusion/exclusion criteria are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 79 years of age, inclusive.
2. Willing and able to give informed consent.
3. Idiopathic RLS, meeting all 4 International RLS Study Group diagnostic criteria.
4. Moderate or severe symptoms, defined as an IRLS score ≥ 15 at screening visit.
5. RLS medications unchanged for 4 weeks prior to baseline.
6. Must have a driver or available transportation (including provided Uber vouchers) to drive them to and from study visits and for other transportation needs during the treatment period.
7. Has a significant other, caregiver, or close acquaintance who knows the subject well and agrees to participate in the subject's neuropsychiatric assessment.
8. Agrees to not take more than 1 gram per day of acetaminophen.
9. Whereas applicable, agrees to utilize an effective method of contraception from screening through at least 4 weeks after the completion of study treatment.

Exclusion Criteria:

1. Secondary RLS, such as Parkinson's disease or end-stage renal disease.
2. Present or past history of another severe sleep disorder.
3. Currently on night shift work schedule.
4. History or diagnosis of schizophrenia, bipolar or a psychotic disorder, severe depression, or any mental health illness that would compromise the safety of the participant.
5. Current suicidal ideation.
6. Severe cognitive impairment (e.g., Alzheimer's Disease, traumatic brain injury).
7. Uncontrolled hypertension.
8. Known or suspected allergy or hypersensitivity to cannabinoids or excipients used in the study drug formulation.
9. Pending legal action or workers compensation.
10. Cannabis use (THC) detectable at the screening/baseline visits.
11. History of drug or alcohol dependence.
12. Use of dopamine blockers, cocaine, or MAO-A inhibitors within 90 days of baseline.
13. Use of any drugs with known interactions with cannabinoids (e.g., tolcapone, clopidogrel, felbamate, warfarin, barbiturates, benzodiazepines, niacin, nicotinamide, isoniazid, ketoconazole, clobazam, valproate, mTOR inhibitors) within 90 days of baseline.
14. Unstable medical condition.
15. Clinically significant laboratory abnormalities.
16. Moderate or severe hepatic impairment.
17. Is pregnant, lactating, or has a positive pregnancy test result pre-dose.
18. Planned elective surgery during study participation.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
To examine the safety and tolerability of oral high CBD extract in idiopathic RLS assessed by frequency of adverse events which will be monitored by patient reported adverse events, vital signs, physical exam, and safety labs during study visits. | Baseline, Visit 3, Visit 4, Visit 5
  Participant reports measures the frequency of adverse events. This will be done with open-ended questions during patient visits and phone calls.
  Abnormal vital signs (BP, HR, RR) at patient visits measures the frequency of participants with adverse events. BP over 130/80 mmHg indicates worse outcomes. Lower scores indicate worse outcomes. HR ranges from 60 to 100 bpm; Scores outside this range indicates worse outcomes. RR ranges from 12-20 bpm. Scores outside this range indicated worse outcomes.
  A neurological exam and routine physical exam will be preformed to examine adverse events. Abnormal findings will constitute as an adverse event.
  Labs (serum CBC w/ diff, serum CMP, urinalysis) will measure frequency of adverse events. Abnormal CBC w/diff, CMP, and urinalysis values will be determined by lab ranges.

SECONDARY OUTCOMES:
To examine the effect of BRC-002 on RLS symptoms assessed through changes from baseline in RLS-6 Severity Scale | Baseline; Day 20
  The RLS-6 Severity Scale ranges from 0-60; increasing scores indicates a worse outcome.
To examine the effect of BRC-002 on RLS symptoms assessed through changes from baseline in change from baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLS) | Baseline; Day 20
  The International Restless Legs Syndrome Study Group Rating Scale (IRLS) measures RLS symptoms. Scores range from 0 to 40, with higher scores indicating a worse outcome.
To examine the effect of BRC-002 on RLS symptoms assessed through changes in sleep quality index (SQI) as measured by the SleepImage Ring | Baseline; Day 20
  The SleepImage Recorder ring measures quality of sleep. Scores range from 0 to 100, with higher scores indicating a better outcome.
To examine the effect of BRC-002 on RLS symptoms assessed through changes in the Pittsburgh Sleep Quality Index (PSQI). | Baseline; Day 20
  The Pittsburg Sleep Quality Index (PSQI) measures sleep quality. Scores range from 0 to 21, with higher scores indicating a worse outcome.
To examine the effect of BRC-002 in sleep measured by change in the Epworth Sleepiness Scale (ESS) | Baseline; Day 20
  The Epworth Sleepiness Scale (ESS)measures daytime sleepiness. Scores range from 0 to 24, with higher scores indicating a worse outcome.
To examine the effect of BRC-002 on RLS symptoms assessed through changes in the Fatigue Severity Scale (FSS). | Baseline; Day 20
  The Fatigue Severity Scale (FSS) measures fatigue. Scores range from 9 to 63, with higher scores indicating a worse outcome.
To examine the effect of BRC-002 in cognition measured by change in the Montreal Cognitive Assessment (MoCA) | Baseline; Day 20
  The Montreal Cognitive Assessment (MoCA) measures cognitive impairment. Scores range from 0 to 30, with higher scores indicating a better outcome.
To examine the effect of BRC-002 in psychiatric symptoms measured by change in the Neuropsychiatric Inventory (NPI) assessment. | Baseline; Day 20
  Neuropsychiatric Inventory (NPI) measures behavior. Scores range from 0 to 144, with higher scores indicating a worse outcome.
To examine the effect of BRC-002 in mood measured by change in the Emotional and Behavioral Dyscontrol Short Form. | Baseline; Day 20
  The Quality of Life in Neurological Disorders Measurement System (Neurol-QOL) measures mood. Scores range from 0 to 100, with higher scores indicating a better outcome.
To examine the effect of BRC-002 on RLS symptoms assessed through changes in Patient Reported Outcome Measurement Information System (PROMIS). | Baseline; Day 20
  Patient Reported Outcome Measurement Information System (PROMIS) measures pain. Scores range from 0 to 100, with higher scores indicating a worse outcome.
To examine the effect of BRC-002 in suicidality measured by change in the Columbia-Suicide Severity Rating Scale (C-SSRS). | Baseline; Day 20
  The C-SSRS measures suicidality in participants. The scores range from 2 through 25; with higher scores indicating worse outcomes.
To examine the effect of BRC-002 on RLS symptoms assessed through changes in Clinical Global Impression (CGI) Scales | Baseline; Day 20
  Clinical Global Impression (CGI) Scales measures improvement in RLS. Scores range from 0 to 7, with higher scores indicating a worse outcome.
To examine the effect of BRC-002 on RLS symptoms assessed through changes in Johns Hopkins Restless Legs Syndrome Quality of Life Questionnaire (RLSQoL). | Baseline; Day 20
  The Johns Hopkins Restless Legs Syndrome Quality of Life Questionnaire (RLSQoL) measures severity of RLS symptoms. Scores range from 0 to 72; with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Bainbridge, Principal Investigator — Skaggs School of Pharmacy

IPD SHARING:
Plan to Share IPD: Yes